CLINICAL TRIAL: NCT05916690
Title: Electrochemotherapy for the Treatment of Vulvar Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institute of Oncology Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERID-KSOPKR-0042/2021
Record Dates: First submitted 2023-06-01; First posted 2023-06-23 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Vulvar Cancer
MeSH Terms: conditions — Vulvar Neoplasms | interventions — Electrochemotherapy; Bleomycin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electrochemotherapy (Experimental)
  Interventions: Drug: Electrochemotherapy with bleomycin or cisplatin

INTERVENTIONS:
Drug: Electrochemotherapy with bleomycin or cisplatin — Combination of drug delivery platform (electroporation) and drug (bleomycin)

SUMMARY:
Electrochemotherapy is a local treatment modality with effectiveness comparable to other local ablation techniques. With electrochemotherapy 80% objective response can be achieved and is suitable for the treatment of different types of tumors. The method is based on increased drug delivery to cells previously exposed to electroporation. The most commonly used cytotoxic agents are bleomycin and cisplatin. The aim of the proposed clinical trial is to determine the efficacy, feasibility and safety of electrochemotherapy in the treatment of vulvar cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Local recurrence of vulvar cancer confirmed by histology
2. The longest diameter of tumor 50 millimeters or less
3. Age more than 18 years
4. Life expectancy of more than 3 months
5. Performance status according to Karnofsky ≥ 70 or < or 2 according to the WHO scale
6. At least 2 weeks have passed since the last treatment
7. The patient must be able to understand the treatment process and possible side effects that may occur during the treatment
8. Signed informed consent form
9. The patient must be presented at a Multidisciplinary Tumor Board

Exclusion Criteria:

1. Life-threatening infection and/or heart failure and/or liver failure and/or markedly impaired pulmonary function and/or other life-threatening systemic diseases
2. Regional or distant metastases
3. Age less than 18 years
4. Major disturbances in the coagulation system (which do not respond to standard therapy - replacement of vitamin K or fresh frozen plasma)
5. Exposure to cumulative bleomycin doses greater than 400 mg
6. Impaired renal function (Creatinine > 150 µmol/L)
7. Epilepsy
8. Pregnancy
9. Patients who are unable to understand the treatment process or refuse to be involved in the treatment process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events 1 month after the treatment | 1 month
  According to CTCAE v5.0
Number of adverse events 2 months after the treatment | 2 months
  According to CTCAE v5.0
Number of adverse events 3 months after the treatment | 3 months
  According to CTCAE v5.0
Number of adverse events 6 months after the treatment | 6 months
  According to CTCAE v5.0
Number of adverse events 9 months after the treatment | 9 months
  According to CTCAE v5.0
Number of adverse events 12 months after the treatment | 12 months
  According to CTCAE v5.0
Response of the tumor to electrochemotherapy according to RECIST criteria | 1 month
  According to RECIST criteria
Response of the tumor to electrochemotherapy according to RECIST criteria | 2 months
  According to RECIST criteria
Response of the tumor to electrochemotherapy according to RECIST criteria | 3 months
  According to RECIST criteria
Response of the tumor to electrochemotherapy according to RECIST criteria | 6 months
  According to RECIST criteria
Response of the tumor to electrochemotherapy according to RECIST criteria | 9 months
  According to RECIST criteria
Response of the tumor to electrochemotherapy according to RECIST criteria | 12 months
  According to RECIST criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Oncology Ljubljana, Ljubljana, Slovenia